CLINICAL TRIAL: NCT00918073
Title: Evaluation of Cardiovascular Effects of Smoking Cessation in HIV Infected Patients
Brief Title: Evaluation of Cardiovascular Effects of Smoking Cessation in HIV Patients
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Tanvir K. Bell, MD, Associate Professor, The University of Texas Health Science Center, Houston
Other Study IDs: UT-GCRC CIMT HIV smokers
Record Dates: First submitted 2009-06-09; First posted 2009-06-11 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-05

CONDITIONS: HIV Infections; Smokers
Keywords: HIV infected smokers; HIV
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIV positive smokers: 50 HIV infected patients who enroll in a parent protocol to quit smoking and elect to participate in this sub-study.

SUMMARY:
We will conduct a sub-study of "An Innovative Telephone Intervention for HIV+ Smokers," (NCT00502827) conducted by Drs. Gritz, Vidrine, and others. This is a randomized, prospective trial that will evaluate a cellular phone delivered counseling intervention versus standard of care for smoking cessation. In our sub-study, we will evaluate rates of progression in atherosclerosis in HIV/AIDS patients who quit smoking versus those who continue smoking by measuring carotid intima-media thickness(CIMT) and biomarkers of atherosclerosis at time point baseline, 1 year, and 3 year. The biomarkers measured include high-sensitivity Creactive protein, homocysteine, and IL-6. We will also evaluate rates of progression of CIMT in those who quit smoking versus those who continue smoking, based on race, sex, state of HIV disease, comorbid diseases, and lipid profile.

DETAILED DESCRIPTION:
HIV/AIDS patients may have an increased risk of myocardial infarction. Traditional risk factors for coronary artery disease, including cigarette smoking, likely play a large role. The prevalence of smoking in the HIV patient population is higher than the general population. We will conduct a sub-study of "An Innovative Telephone Intervention for HIV+ Smokers," (NCT00502827) conducted by Drs. Gritz, Vidrine, and others. This is a randomized prospective trial that will evaluate a cellular phone delivered counseling intervention versus standard of care for smoking cessation. In our sub-study, we will evaluate rates of progression in atherosclerosis in HIV/AIDS patients who quit smoking versus those who continue smoking by measuring carotid intima-media thickness(CIMT) and biomarkers of atherosclerosis at time point baseline, 1 year, and 3 year. The biomarkers measured include high-sensitivity Creactive protein, homocysteine, and IL-6. We will also evaluate rates of progression of CIMT in those who quit smoking versus those who continue smoking based on race, sex, state of HIV disease, comorbid diseases and lipid profile. The central hypothesis is that smoking cessation win slow the atherosclerosis progression in HIV patients. A successful behavioral intervention is being evaluated in the parent study. The goal of this sub-study is to assess the effect of a modifiable coronary artery disease risk factor, smoking, in HIV/AIDS patients through this collaboration of cardiovascular expertise and metrics.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet eligibility criteria for "An innovative telephone intervention for HIV-positive smokers".
* Patients who consent to the sub-study.
* Patients who are able to participate in the study for 3 years.

Exclusion Criteria:

* Patients with a history of coronary bypass surgery, percutaneous coronary intervention, valve replacement, pacemaker or defibrillator implantation.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HIV positive smokers who enroll in a smoking cessation trial who elect to participate in this substudy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2007-11; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will compare change in mean maximum carotid IMT over the course of the study between HIV patients who quit smoking and those that continue to smoke. | 3 years

SECONDARY OUTCOMES:
The secondary endpoint will evaluate change in mean carotid IMT. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Tanvir K Bell, MD, Principal Investigator — UT Health Science Center, Houston
Locations (1):
- Thomas Street Health Center, Houston, Texas, United States